CLINICAL TRIAL: NCT02650245
Title: Breath and Blood Ammonia Response to an Oral Protein Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr. Steve Solga, M.D., St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-59
Record Dates: First submitted 2015-10-15; First posted 2016-01-08 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Cirrhosis
Keywords: breath; gastroenterology; ammonia; blood; protein; cirrhosis; encephalopathy
MeSH Terms: conditions — Fibrosis; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate protein and 10gm lactulose (Experimental): 40% of daily recommended intake of protein based on weight
  Interventions: Dietary Supplement: EAS Myoplex Protein Drink + 10gm lactulose

INTERVENTIONS:
Dietary Supplement: EAS Myoplex Protein Drink + 10gm lactulose

SUMMARY:
The investigators specific aim is to evaluate the changes in breath ammonia in comparison to blood ammonia and other physiologic markers after a moderate oral protein challenge in healthy subjects and subjects with liver cirrhosis.

DETAILED DESCRIPTION:
Ammonia is an important molecule relevant to numerous diseases, especially to the millions of patients with cirrhosis worldwide. Venous blood ammonia via limb phlebotomy, can at best roughly estimate whole body ammonia, but says little or nothing about intestinal production, and cannot "source" ammonia to any particular organ or body compartment. Unfortunately, there are no presently available better tests. Therefore, despite these acknowledged limitations, venous ammonia the "bronze standard" benchmark by which new metrics are assessed.

The present protocol attempts to address both concerns and build upon the investigators prior high protein experience. By using a standard moderate protein challenge, the investigators can evaluate the breath ammonia responsiveness in healthy subjects and those with cirrhosis. This protocol leverages the power of breath research to evaluate responses to oral challenges. This remains a key asset of breath research.

Since the protocol proposes a moderate protein challenge, the investigators can evaluate disease states with minimal or no risk. As with past high protein studies, lactulose (10gm) will still be added to provoke a hydrogen response.

ELIGIBILITY:
Inclusion Criteria:

* <18 and <75 yrs of age

Exclusion Criteria:

* Diabetic, smoker, substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Levels of Ammonia (parts per billion) in response to an oral protein challenge using the Bedfont breath monitor | 5 hours
  Evaluating change in breath ammonia at hour 5 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Steve Solga, M.D., Principal Investigator — St. Luke's University Hospital and Health Network
Locations (1):
- St. Luke's University Hospital and Health Network, Bethlehem, Pennsylvania, United States